CLINICAL TRIAL: NCT01757613
Title: Three-armed, Randomized, Double-blind Dose-finding Trial on Efficiency and Safety of AK 3012 in 3 Different Concentrations in Patients With Actinic Keratosis Olsen Grade I/II
Brief Title: Study Whose Purpose is to Find an Optimal Dose for the Treatment With AK 3012 in Patients With Actinic Keratosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dolorgiet GmbH & Co. KG (Industry)
Collaborators: CenTrial GmbH (Industry); d.s.h. statistical services GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KER-001; 2012-002529-30 (EudraCT Number)
Record Dates: First submitted 2012-12-18; First posted 2012-12-31 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Actinic Keratosis Olsen Grade I/II

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- AK 3012 a for topical use (Active Comparator)
  Interventions: Drug: AK 3012
- AK 3012 b for topical use (Active Comparator)
  Interventions: Drug: AK 3012
- AK 3012 c for topical use (Active Comparator)
  Interventions: Drug: AK 3012

INTERVENTIONS:
Drug: AK 3012 — cutaneous use twice a day

SUMMARY:
In this three-armed dose-finding trial 3 AK 3012 topical formulations shall be investigated with respect to safety and efficacy in order to identify the optimal concentration in the topical formulation.

The main objective of the trial is to determine the optimal concentration of the active agent in the topical formulation as quantified by the change of the number of skin alterations in pre-defined areas in a time period from inclusion in the trial until the end of treatment (3 months) or prior complete healing.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years
* Gender: male and female
* Actinic Keratosis (Olsen grade I/II)
* at least 5 actinic keratoses on the scalp, forehead, face, extremities, and/ or decollete
* no treatment of the actinic keratoses within the previous 3 months before inclusion in the study
* histologic confirmation of the diagnosis actinic keratosis by biopsy
* good general condition
* normal laboratory values (creatinine, urea, Glutamate-Oxalacetate Transaminase (GOT),Glutamate-Pyruvate Transaminase (GPT), gamma-glutamyl transferase (GGT), Lactate dehydrogenase (LDH)) and blood count at study start not higher than 1.5 x upper norm limit
* Female patients must be tested negative for pregnancy before inclusion in the trial. During the trial, female patients have to apply a generally accepted form of birth control (i.e. oral estrogen- and gestagen containing contraceptives; estrogen containing skin plaster/ tape, hormone implant, hormone contraceptive coil, sterilisation; sexual abstinence) or being post-menopausal for at least 2 years.
* Willing and able to participate in the screening and all trial specific procedures in compliance with the protocol
* Signed written informed consent

Exclusion Criteria:

* Known allergy against nonsteroidal antiphlogistics and/ or against excipients of the investigational medicinal product
* Presence of immunosuppression
* Treatment with 5-fluorouracil, cyclosporine, retinoids, glycolic acid, imiquimod, trichloroacetic acid during the trial or 12 weeks before inclusion in the trial
* Continuous treatment with nonsteroidal antiphlogistics with the exception of low-dose acetylsalicylic acid (100 mg) for inhibition of thrombocyte aggregation
* Planned treatment with photodynamic therapy during participation in the trial
* Pregnancy or lactation
* Participation in another clinical trial within 3 months before inclusion in the current trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change of skin alterations during treatment period | 90 days: Between Visit 0 (day 0) and Visit 3 (day 90)

SECONDARY OUTCOMES:
Change of visible skin alterations during treatment period | 90 days: Between Visit 0 (day 0) and Visit 3 (day 90)
Tolerability of the investigated medicinal product | 90 days: Between Visit 0 (day 0) and Visit 3 (day 90)
  Tolerability will be assessed on the basis of adverse events
Adverse events | 90 days: Between Visit 0 (day 0) and Visit 3 (day 90)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Yazdi, Dr. med, Principal Investigator — Eberhard-Karls-Universität Tübingen; Angelika Trapp, Study Director — Dolorgiet GmbH & Co. KG
Locations (7):
- Germany (7):
  - Blaubeuren Abbey
  - Friedrichshafen
  - Hamburg
  - Langenau
  - Radolfzell
  - Stuttgart
  - Tübingen